CLINICAL TRIAL: NCT02620410
Title: Treatment of REfractory Overactive BLadder With the AXonics Sacral Neuromodulation System (RELAX-OAB)
Acronym: RELAX-OAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Axonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105-0010
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Overactive Bladder
Keywords: OAB
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Axonics SNM System (Other): Axonics SNM Therapy for urinary control is indicated for the treatment of urinary retention and the symptoms of overactive bladder, including urinary urge incontinence and significant symptoms of urgency-frequency alone or in combination, in patients who have failed or could not tolerate more conservative treatments.
  Interventions: Device: Axonics Sacral Neuromodulation (SNM) System

INTERVENTIONS:
Device: Axonics Sacral Neuromodulation (SNM) System — The implantable components of the Axonics Sacral Neuromodulation (SNM) System consist of an IPG and tined lead. Additional components include a clinician programmer, surgical tool kit, recharging kit, and patient remote control.
  Other Names: Axonics SNM System

SUMMARY:
The RELAX-OAB (Treatment of REfractory Overactive BLadder with the AXonics Sacral Neuromodulation System) is a post-market clinical follow-up (PMCF) study designed to confirm the performance of the Axonics Sacral Neuromodulation (SNM) System as an aid in the treatment of the symptoms of overactive bladder (OAB) as well as capturing patient satisfaction and quality of life data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OAB as demonstrated on a 3-day voiding diary defined as ≥ 8 voids/day, and/or a minimum of 2 involuntary leaking episodes in a 72-hour period
* Positive motor response on at least two implanted electrodes during intraoperative test
* Failed, or are not a candidate for more conservative treatment (e.g., pelvic floor training, biofeedback, behavioral modification, oral pharmacotherapy)
* No changes to current regimen of medications that affect bladder function for at least 4 weeks prior to beginning the baseline voiding diary
* Willing and capable of providing informed consent
* Capable of participating in all testing associated with this clinical investigation

Exclusion Criteria:

* Primary stress incontinence or mixed incontinence where the stress component overrides the urgency component
* Current urinary tract mechanical obstruction such as benign prostatic enlargement or urethral stricture
* Interstitial cystitis or bladder pain syndrome as defined by either AUA or EAU guidelines
* History of any pelvic cancer
* Any significant medical condition that is likely to interfere with study procedures, device operation, or likely to confound evaluation of study endpoints
* Any psychiatric or personality disorder at the discretion of the study physician
* PHQ-9 Patient Depression Score ≥ 10
* Current symptomatic urinary tract infection (UTI) or more than 3 UTIs in past year
* Any neurological condition that may interfere with normal bladder function, including stroke, multiple sclerosis, Parkinson's disease, clinically significant peripheral neuropathy, or spinal cord injury (e.g., paraplegia)
* Severe or uncontrolled diabetes (A1C > 8, documented in the last 3 months) or diabetes with peripheral nerve involvement
* Treatment of urinary symptoms with botulinum toxin therapy in the past 12 months
* Treatment of urinary symptoms with tibial nerve stimulation in the past 3 months
* Previously implanted with a sacral neuromodulation device or participated in a sacral neuromodulation trial
* Subject with a documented history of allergic response to titanium, zirconia, polyurethane, epoxy, or silicone
* Knowledge of planned MRIs, diathermy, or high output ultrasonic exposure
* Any other active implanted devices including neurostimulators (e.g., cochlear implant, pacemaker) and/or drug delivery pumps, whether turned on or off
* Passive implants (e.g., prostheses) are allowed, but no implanted metal should be at the Neurostimulator implant site
* A female who is breastfeeding or of child-bearing potential with a positive urine pregnancy test or not using adequate contraception
* Participation in a current clinical trial or within the preceding 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Mean change in ICIQ-OABqol HRQL Total Score compared to baseline. | 3 Months
  A disease-specific quality of life questionnaire. The ICIQ-OABqol is a psychometrically robust patient-completed questionnaire evaluating quality of life (QoL) in patients with overactive bladder for use in research and clinical practice across the world. The ICIQ-OABqol is the OAB-q adapted for use within the ICIQ structure and provides a detailed and robust measure to assess the impact of overactive bladder on quality of life. It is an ideal research tool as it explores in detail the impact on patients' lives of overactive bladder. The Third International Consultation on Incontinence recommended that all randomised trials evaluating treatments for incontinence use high quality questionnaires, in particular the ICIQ, to assess impact on patient outcome and facilitate comparisons. The ICIQ-OABqol provides a robust measure for this purpose.

SECONDARY OUTCOMES:
Rate of serious adverse device effects (SADEs) | 3 Months, 1 Year, 2 Year post-implantation
Rate of adverse device effects (ADEs) | 3 Months, 1 Year, 2 Year post-implantation
Rate of adverse procedure effects (APEs) | 3 Months, 1 Year, 2 Year post-implantation
Rate of serious adverse events (SAEs) | 3 Months, 1 Year, 2 Year post-implantation
Rate of adverse events (AEs) | 3 Months, 1 Year, 2 Year post-implantation
Device performance metrics | 3 Months, 1 Year, 2 Year post-implantation
  Data recorded from the patient's devices (Device Readings)
Average leaks per day (3-day voiding diary) | 3 Months, 1 Year, 2 Year post-implantation
Average voids per day (3-day voiding diary) | 3 Months, 1 Year, 2 Year post-implantation
Percent of subjects with successful treatment | 3 Months, 1 Year, 2 Year post-implantation
  Defined as either 1) a 50% improvement in the number of average leaks or the number of voids per day or 2) a return to a normal number of voids per day (<8 voids)
SF-12 | 3 Months, 1 Year, 2 Year post-implantation
  General quality of life questionnaire
EQ-5D | 3 Months, 1 Year, 2 Year post-implantation
  Questionnaire assessing general quality of life
ICIQ-UI Short Form | 3 Months, 1 Year, 2 Year post-implantation
  Quality of life questionnaire assessing urinary incontinence
ICIQ-OABqol | 3 Months, 1 Year, 2 Year post-implantation
  Quality of life questionnaire assessing over active bladder
I-QOL | 3 Months, 1 Year, 2 Year post-implantation
  Quality of life questionnaire assessing urinary incontinence
Patient satisfaction with treatment | 3 Months, 1 Year, 2 Year post-implantation
  Questionnaire in scale format assessing treatment-specific satisfaction
Healthcare utilization | 3 Months, 1 Year, 2 Year post-implantation
  Questionnaire about subject's medical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sohier Elneil, MRCOG, PhD, Principal Investigator — University College London Hospital & National Hospital for Neurology & Neurosurgery
Locations (6):
- UZ Leuven, Leuven, Belgium
- France (2):
  - Hospices Civils de Lyon, Lyon
  - Chu De Nantes - Hôtel-Dieu, Nantes
- Netherlands (2):
  - Maastricht University Medical Center, Maastricht
  - Erasmus Medical Center, Rotterdam
- University College London Hospital, London, United Kingdom